CLINICAL TRIAL: NCT02251821
Title: JAK Inhibitor Prior to Allogeneic Stem Cell Transplant for Patients With Primary and Secondary Myelofibrosis: A Prospective Study
Brief Title: JAK Inhibitor Before Donor Stem Cell Transplant in Treating Patients With Primary or Secondary Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rachel Salit, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9033; NCI-2014-01882 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9033 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9214017 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-09-12; First posted 2014-09-29 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Busulfan; Cyclophosphamide; fludarabine phosphate; Melphalan; Methotrexate; merphos; Mycophenolic Acid; ruxolitinib; Tacrolimus; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib, transplant) (Experimental): Patients receive a ruxolitinib and undergo myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis; see detailed description.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Methotrexate; Drug: Mycophenolate Mofetil; Drug: Ruxolitinib; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424; Jakafi
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation; SCT_TBI
Procedure: Umbilical Cord Blood Transplantation — Undergo umbilical cord blood transplant
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase II trial studies how well giving a JAK inhibitor before a donor stem cell transplant works in treating patients with myelofibrosis that developed without another condition (primary) or evolved from other bone marrow disorders (secondary). JAK inhibitors are a class of drugs that may stop the growth of abnormal cells by blocking an enzyme needed for cell growth. Giving a JAK inhibitor such as ruxolitinib before a donor stem cell transplant may help reduce symptoms of myelofibrosis such as inflammation and enlargement of the spleen, improve the patient's general physical condition, and prevent complications from occurring after the transplant. Infusing healthy stem cells from a donor into the patient may help the patient's bone marrow work normally and make stem cells, red blood cells, white blood cells, and platelets. Giving a JAK inhibitor before a donor stem cell transplant may help improve transplant outcomes in patients with myelofibrosis.

DETAILED DESCRIPTION:
OUTLINE:

PART 1: Patients receive ruxolitinib orally (PO) twice daily (BID) from at least 8 weeks prior to the start of conditioning through day -4 before transplantation, with a taper schedule reducing the dose every 2-3 days beginning after day -4.

PART 2: Patients are assigned to 1 of 2 conditioning regimens at the discretion of the clinical provider and Clinical Coordinators Office (CCO).

MYELOABLATIVE CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -8 to -6 (umbilical cord blood transplant recipients only), cyclophosphamide IV on days -7 and -6, and busulfan IV over 3 hours on days -5 to -2.

REDUCED-INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and melphalan IV over 15-30 minutes on days -3 and -2. Patients also undergo total-body irradiation (TBI) on day -1 (umbilical cord blood transplant recipients only).

TRANSPLANT: Patients undergo allogeneic hematopoietic stem cell transplant or umbilical cord blood transplant on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive tacrolimus IV continuously (inpatients) or over 1-2 hours twice daily (BID) (outpatients) or orally (PO) BID on days -1 to +180 (patients receiving related or unrelated stem cells) or days -3 to +180 (patients receiving umbilical cord blood) with taper beginning on day +56 (related donor recipients) or +100 (unrelated donor or umbilical cord blood recipients) in the absence of GVHD. Patients also receive methotrexate IV on days +1, +3, +6, and +11 (related and unrelated donor recipients only) or mycophenolate mofetil IV or PO every 8 hours on days 0 to +40 with taper to day +96 (umbilical cord blood transplant recipients only).

After completion of study treatment, patients are followed up at 6 months, 1 year, and then yearly for 4 years.

ELIGIBILITY:
Inclusion Criteria:

PART 1:

* PART 1: Disease criteria

  * Diagnosis of primary MF (PMF) as defined by the 2008 World Health Organization classification system or diagnosis of secondary MF as defined by the International Working Group (IWG) for Myeloproliferative Neoplasms Research and Treatment criteria
  * Patients meeting the criteria for intermediate-1, intermediate-2 or high-risk disease by the Dynamic International Prognostic Scoring System (DIPSS) or DIPSS-plus scoring system
* PART 1: Ability to understand and the willingness to sign a written informed consent document
* PART 1: Patient must be a potential hematopoietic stem cell transplant candidate

PART 2:

* PART 2: Meeting criteria for 1st phase as above, at time of initiation of JAK inhibitor, including ability to understand and willingness to sign a written informed consent; patients arriving to our institution for transplant and not enrolled in Part 1 may still be enrolled in Part 2 if Part 1 criteria met; these patients will have Part 1 endpoints transcribed from medical records
* PART 2: Received ruxolitinib for at least 8 weeks immediately prior to conditioning and be able to continue until Day -4 pre-transplant
* PART 2: Performance status score

  * Karnofsky >= 70
* PART 2: Calculated creatinine clearance using the Cockcroft-Gault formula or 24 hr urine creatinine clearance must be > 60 ml/min
* PART 2: Total serum bilirubin must be < 3 mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* PART 2: Transaminases must be < 3 x the upper limit of normal
* PART 2: Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* PART 2: Diffusing capacity of the lung for carbon monoxide (DLCO) corrected > 60% normal

  * May not be on supplemental oxygen
* PART 2: Left ventricular ejection fraction > 40% OR
* PART 2: Shortening fraction > 26%
* PART 2: Comorbidity Index < 5 at the time of pre-transplant evaluation

DONOR:

* DONOR: Human leukocyte antigen (HLA)-matched or 1 antigen mismatched sibling donor
* DONOR: 10 of 10 HLA-matched or 1 allele mismatched (9 of 10) unrelated donor
* DONOR: Peripheral blood is preferred over bone marrow for non-umbilical cord blood recipients
* DONOR: Umbilical cord blood units will be selected according to the following umbilical cord blood graft selection criteria; one or 2 cord blood (CB) units may be used to achieve the required cell dose
* DONOR: The CB graft(s) must be matched at 4-6 HLA-A, B, DR Beta 1 (DRB1) loci with the recipient and therefore may include 0-2 mismatches at the A or B or DRB1 loci; unit selection will be based on cryopreserved nucleated cell dose and intermediate resolution A, B antigen and DRB1 allele typing for determination of HLA-match; while HLA-C antigen/allele level typing is not considered in the matching criteria, if available, it may be used to optimize unit selection
* DONOR: Selection of two CB units is allowed to provide sufficient cell dose (see below for algorithm to determine single versus double unit transplant); when multiple units are selected, the following rules apply:

  * The CB unit with the least HLA disparity (with the patient) will be selected first (i.e., selection priority is 6/6 match > 5/6 match > 4/6 match); additional CB units then may be selected to achieve the required cell dose, as outlined below; if a second unit is required, this unit will be the unit that most closely HLA matches the patient and meets minimum size criteria outlined below of at least 1.5 x 10^7 total nucleated cells (TNC)/kg (i.e. a smaller, more closely matched unit will be selected over a larger, less well matched unit as long as minimum criteria are met)
  * If two CB units are used:

    * The total cell dose of the combined units must be at least 3.0 x 10^7 TNC per kilogram recipient weight
    * Each CB unit MUST contain at least 1.5 x 10^7 TNC per kilogram recipient weight
  * Algorithm for determining single versus double unit cord blood transplant:

    * Match grade 6/6: TNC dose >= 2.5 x 10^7/kg
    * Match grade 5/6, 4/6: TNC dose >= 4.0 (+/- 0.5) x 10^7/kg
* DONOR: General comments:

  * Units will be selected first based on the TNC dose and HLA matching
  * Cluster of differentiation (CD)34+ cell dose will not be used for unit selection unless 2 units of equal HLA-match grade are available; in this case, the unit with the larger CD34+ cell dose (if data available) should be selected
  * A CB unit that is 5/6 mismatched but homozygous at the locus of mismatch should be chosen over a 5/6 unit with bidirectional mismatch even if the latter unit is larger (has more cells); this also applies to 4/6 units; this is only applicable to choosing units within a given match grade
  * Other factors to be considered:

    * Within the same HLA match grade, matching at DR takes preference
    * Cord blood banks located in the United States are preferred
  * Up to 5% of the cord blood product(s), when ready for infusion, may be withheld for research purposes as long as thresholds for infused TNC dose are met; these products will be used to conduct studies involving the kinetics of engraftment and immunobiology of double cord transplantation

Exclusion Criteria:

PART 1:

* PART 1: Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* PART 1: Uncontrolled viral, bacterial, or fungal infections at the time of study enrollment
* PART 1: History of prior allogeneic transplant
* PART 1: Pregnant or breastfeeding (only if patients have not been started on ruxolitinib [Rux] by their primary oncologist prior to enrollment)

PART 2:

* PART 2: Uncontrolled viral or bacterial infection at the time of study enrollment
* PART 2: Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* PART 2: History of HIV infection
* PART 2: Pregnant or breastfeeding
* PART 2: Patients without an HLA-identical or 1-allele-mismatched related donor or unrelated donor or umbilical cord blood units that meet transplant criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2025-12-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Salit, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original accrual goal to reach the primary endpoint was 48 patients. An additional 15 patients were added in order to collect samples for our translational work on GVHD biomarkers (total 63). We stopped our accrual at 61 patients when we opened our current study looking giving Rux in the peri-transplant setting.
Groups:
- Treatment (ruxolitinib, transplant): Patients receive a ruxolitinib and underwent a myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis; see detailed description.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic hematopoietic stem cell transplant
  Busulfan: Given IV
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Melphalan: Given IV
  Methotrexate: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Ruxolitinib: Given PO
  Tacrolimus: Given IV or PO
  Total-Body Irradiation: Undergo TBI
  Umbilical Cord Blood Transplantation: Undergo umbilical cord blood transplant
Period: Overall Study
Arm/Group | Treatment (ruxolitinib, transplant)
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All transplanted patients
Groups:
- Treatment (Ruxolitinib, Transplant): Patients receive a ruxolitinib for at least 8 weeks and undergo myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis; see detailed description.
Arm/Group | Treatment (Ruxolitinib, Transplant)
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 57
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance Status (KPS) at time of HCT [Count of Participants; unit: Participants] — "Karnofsky performance scale was used for rating participant activities of daily living. It rated participant on 11-step scale ranged from 0-100, higher score=participant is better able to carry out daily activities. The lower the score, the worse the survival for most serious illnesses.
  Participants
    100 | 10
    90 | 28
    80 | 19
    70 | 4
DIPSS (Dynamic International Prognostic Scoring System) for Myelofibrosis [Count of Participants; unit: Participants] — Age, years. ≤650. >65+1. White blood cell count, x10⁹/dL. ≤250. >25+1. Hemoglobin, g/dL. ≥100. <10+2. Peripheral blood blasts. <1%0. ≥1%+1. Constitutional symptoms. No0. Yes+1.
  The DIPSS assigns two, rather than one, adverse points for hemoglobin <10 g/dL, and the risk categorization is accordingly modified: low (0 adverse points), intermediate-1 (1 or 2 points), intermediate-2 (3 or 4 points) and high (5 or 6 points). A higher score is a worse prognosis.
  Participants
    Low-risk | 2
    Intermediate 1 risk | 16
    Intermediate 2 risk | 41
    High-risk | 2
Donor Source [Count of Participants; unit: Participants]
  HLA-matched sibling | 25
  Matched unrelated | 26
  Cord Blood | 6
  1 allele mismatched unrelated | 4
Conditioning Regimen Intensity [Count of Participants; unit: Participants]
  High Intensity Myeloablative | 41
  Reduced Intensity Myeloablative | 20
Primary or Secondary Myelofibrosis [Count of Participants; unit: Participants]
  Primary MF | 36
  Secondary MF | 25

OUTCOME MEASURES:

1. Primary Outcome: 2-year Overall Survival (OS) in Patients With Myelofibrosis (MF) Who Receive Treatment With a JAK Inhibitor Followed by an Allogeneic Transplant
Description: OS was defined as the time from date of transplantation to date of death due to any cause. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. The 2-year survival probability was estimated using the Kaplan-Meier method and a 2-sided 95% confidence interval (CI).
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treatment (ruxolitinib, transplant): Patients receive a ruxolitinib and undergo myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percentage of participants | 78.24 [68.43 to 89.45]

2. Secondary Outcome: Percentage of Participants With Acute Graft Versus Host Disease (GVHD) Grade II-IV
Description: Percentage of Participants with Grade II-IV acute GVHD in the first 100 days post HCT.
Time Frame: Up to 100 days post-transplant
Population: Only 58 of the 61 patients had acute GVHD scoring completed
Measure: Number; unit: percent of participants
Groups:
- Treatment (ruxolitinib, transplant): Patients receive a ruxolitinib and underwent a myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis;
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 58
percent of participants | 68.97

3. Secondary Outcome: Percentage of Participants With Chronic Graft Versus Host Disease (GVHD)
Description: Max grade of chronic GVHD mild, moderate or severe at any time within the first 2 years following transplant.
Time Frame: 2 years
Measure: Number; unit: percent of participants
Groups:
- Treatment (ruxolitinib, transplant): Patients receive a ruxolitinib and underwent a myeloablative or reduced-intensity conditioning followed by transplant and GVHD prophylaxis.
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percent of participants | 60.66

4. Secondary Outcome: Percentage of Patients Who Had Relapsed Disease at 1 Year
Description: Patients who had evidence of residual disease by molecular, flow cytometric or cytogenetics/FISH were considered relapsed disease.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percent of participants | 8.29 [3.02 to 17]

5. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Patients who died in remission between day of transplant and day 100.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percent of participants | 4.92 [1.28 to 12.47]

6. Secondary Outcome: Non-relapse Mortality (NRM)
Time Frame: 1 year
Measure: Number (90% Confidence Interval); unit: percent of participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percent of participants | 13.26 [6.15 to 23.15]

7. Secondary Outcome: Number of Patients Who Experienced Primary Graft Failure/Rejection
Description: Patients who failed to achieve ANC > 500 x 3 or chimerism > 5% by day 42 post-transplant.
Time Frame: Up to 42 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
Participants | 1

8. Secondary Outcome: Number of Patients Who Experienced Secondary Graft Failure/Poor Graft Function
Description: Patients who engrafted with an ANC >500 x 3 or chimerism > 5% and then became neutropenic with ANC <500x3 days or chimerism <5% without evidence of relapse.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
Participants | 2

9. Secondary Outcome: Percentage of Patients With a Max Grade of Moderate and Severe Chronic GVHD at Any Time Before 2 Years Post Transplant.
Description: Includes patients who had a max grade of moderate or severe chronic GVHD by the NIH scoring system at any time between day 0 and 2 years post transplant.
Time Frame: 2 years post-HCT
Measure: Number; unit: percent of participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 61
percent of participants | 44.26

10. Secondary Outcome: Percentage of Participants With Acute Graft Versus Host Disease Grade III-IV GVHD
Description: Patients who had a max grade of III-IV acute GVHD any time between Day 0 and Day 100.
Time Frame: 100 days
Population: Only 58 of the 61 patients had acute GVHD scoring completed
Measure: Number; unit: percent of participants
Arm/Group | Treatment (ruxolitinib, transplant)
Number analyzed (Participants) | 58
percent of participants | 17.24

ADVERSE EVENTS:
Time Frame: Serious AEs and other AEs were assessed for up to 100 days. All-Cause Mortality assessed for up to 5 years.
Description: See attached protocol
Groups:
- Treatment (ruxolitinib, transplant): Patients receive a ruxolitinib and underwent a myeloablative or reduced-intensity conditioning followed by transplant and calcineurin inhibitor based GVHD prophylaxis.
Arm/Group | Treatment (ruxolitinib, transplant)
All-Cause Mortality (participants affected / at risk) | 14/61
Serious Adverse Events (participants affected / at risk) | 7/61
Other Adverse Events (participants affected / at risk) | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ruxolitinib, transplant) (N=61)
Sepsis (Infections and infestations) | 1 (1)
Infections Viral (Infections and infestations) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (ruxolitinib, transplant) (N=61)
Febrile Neutropenia (Blood and lymphatic system disorders) | 27 (27)
Hypocellular Marrow (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Infections-Bacterial (Infections and infestations) | 30 (30)
Infections Viral (Infections and infestations) | 18 (18)
Infections Fungal (Infections and infestations) | 4 (4)
Infections Other (Infections and infestations) | 6 (6)
Elevated Troponin (Cardiac disorders) | 1 (1)
Arrythmia (Cardiac disorders) | 4 (4)
tachycardia (Cardiac disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 39 (39)
Nausea (Gastrointestinal disorders) | 12 (12)
Vomiting (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Abdominal Distention (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 10 (10)
Colitis (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Abdominal (Gastrointestinal disorders) | 2 (2)
Hemorrhage (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Pneumatosis Intestinalis (Gastrointestinal disorders) | 1 (1)
Neutropenic Enterocolitis (Gastrointestinal disorders) | 1 (1)
Anasarca (General disorders) | 1 (1)
sinusoidal outlet obstruction (Hepatobiliary disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 2 (2)
elevated total bilirubin (Hepatobiliary disorders) | 9 (9)
Elevated ALT (Hepatobiliary disorders) | 6 (6)
Elevated AST (Hepatobiliary disorders) | 1 (1)
Serum Creatinine Increased (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Pain-Lumbosacral (Musculoskeletal and connective tissue disorders) | 1 (1)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1)
Weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
altered mental status (Psychiatric disorders) | 3 (3)
anxiety (Psychiatric disorders) | 2 (2)
psychosis (Psychiatric disorders) | 1 (1)
cystitis-non infectious (Renal and urinary disorders) | 1 (1)
viral cystitis (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
toxic erythema (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (3)
blisters (Skin and subcutaneous tissue disorders) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
hypotension (Vascular disorders) | 2 (2)
hypertension (Vascular disorders) | 3 (3)
right atrial thrombus (Vascular disorders) | 1 (1)
ventral hernia (Injury, poisoning and procedural complications) | 1 (1)
hemorrhagic pituitary mass (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02251821/Prot_SAP_000.pdf